CLINICAL TRIAL: NCT00867477
Title: A Biomarker Study Comparing the Pulmonary Metabolic Radiation Response Versus Exhaled Nitric Oxide in Patients Who Receive Thoracic Radiotherapy
Brief Title: PMRR-NO: Pulmonary Metabolic Radiation Response Versus Exhaled Nitric Oxide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008-0632
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Gastrointestinal Disease; Esophageal Cancer; Lung Cancer
Keywords: Cancer of esophagus; Gastrointestine; esophagus cancer; Positron emission tomography; PET scan; Nitric oxide; NO; NO Breathing Test; Respiratory symptoms questionnaire
MeSH Terms: conditions — Gastrointestinal Diseases; Esophageal Neoplasms; Lung Neoplasms | interventions — Surveys and Questionnaires; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Esophagus Cancer (Experimental): Breathing Test + Respiratory Symptoms Questionnaire
  Interventions: Procedure: Breathing Test; Behavioral: Respiratory Symptoms Questionnaire
- Cohort 2: Lung Cancer (Experimental): Breathing Test + Respiratory Symptoms Questionnaire
  Interventions: Procedure: Breathing Test; Behavioral: Respiratory Symptoms Questionnaire; Procedure: Pet Scan

INTERVENTIONS:
Procedure: Breathing Test — Exhale into NO breath analyzer for 10 seconds, repeated 3 times (before radiation therapy starts, after completing radiation therapy, and after scheduled PET scan).
Behavioral: Respiratory Symptoms Questionnaire — 3 page questionnaire about breathing and any symptoms experienced, at each of 2 NO breathing tests.
  Other Names: survey
Procedure: Pet Scan — Between 40 and 50 days after the end of the radiation therapy. Ten (10) participants will receive a second PET scan within 2-7 days after the first PET scan in order to check reproducibility.
  Arms: Cohort 2: Lung Cancer

SUMMARY:
The goal of this clinical research study is to use a new breathing test that measures the amount of nitric oxide (NO) you exhale. Researchers want to compare your "NO" levels to the amount of inflammation in your lungs, as measured using a positron emission tomography (PET) scan reading, and with respiratory symptoms questionnaire.

DETAILED DESCRIPTION:
Lung Cancer Cohort:

NO Breathing Test:

If you agree to take part in this study, you will have a breathing test performed before starting radiation therapy, weekly during radiation therapy and, about 6 weeks after the end of radiation therapy on the same day of your restaging PET scan. The breathing test measures how much NO you exhale while breathing. To complete this test, you will exhale into a device called an "NO breath analyzer" for 10 seconds. You will repeat this test 3 times. The results of this test will give researchers information about possible inflammation in your lungs. The results of this test will be compared to the results of your PET scan.

For the first exhaled NO testing session, and any session in which you produce a high enough NO level, you will have the NO breath test repeated up to 4 times. The staff will ask you to exhale at different speeds during these repeated sessions, in order to learn where in your lungs the NO is coming from.

Respiratory Symptoms Questionnaire:

At each visit when you have NO breathing tests, you will be asked to complete a questionnaire about your breathing and any symptoms you may be having. A research assistant will be able to help you with completing the questionnaire. It should take about 10 minutes to complete the questionnaire.

PET scans:

After completing your radiation therapy, you will receive a PET scan as part of this study. The PET scan will be scheduled for you between 40 and 50 days after the end of the radiation therapy. A study staff member will call you with the PET scan date. Ten (10) participants will receive a second PET scan within 2-7 days after the first PET scan in order to check reproducibility.

For up to 6 hours before the PET scan, you must not eat or drink anything except water. A small tube will be placed in your arm, and you will receive an injection of a very small amount of a mildly radioactive sugar material into your bloodstream. The radioactive nature of this injected material allows the scanner to "see" it in certain places in your body. After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for between 45 and 90 minutes. During the scan, you will lie flat on your back on a table. The scan itself may last up to 1 hour.

Length of Study:

You will remain on study for up to 7 months. After you have completed the breathing tests, blood draws, questionnaires, and PET scans, your participation on this study will be over.

This is an investigational study. The device (called an NO breath analyzer) used in this study is FDA approved and commercially available for measuring exhaled NO levels in patients with asthma. The use of the PET scan and blood test to check lung inflammation is also investigational.

Up to 150 patients (up to 47 with lung cancer) will take part in this study. All will be enrolled at MD Anderson.

Esophageal Cancer Cohort:

NO Breathing Test:

If you agree to take part in this study, you will have a breathing test performed before starting radiation therapy, about 5 weeks later after radiation therapy is complete (at the end of radiation therapy), and the same day of your restaging PET scan. The breathing test measures how much NO you exhale while breathing. To complete this test, you will exhale into a device called an "NO breath analyzer" for 10 seconds. You will repeat this test 3 times. The results of this test will give researchers information about possible inflammation in your lungs. The results of this test will be compared to the results of your PET scan.

For the first exhaled NO testing session, and any session in which you produce a high enough NO level, you will have the NO breath test repeated up to 4 times. The staff will ask you to exhale at different speeds during these repeated sessions, in order to learn where in your lungs the NO is coming from.

Respiratory Symptoms Questionnaire:

At each visit when you have 3 NO breathing tests, you will be asked to complete a questionnaire about your breathing and any symptoms you may be having. A research assistant will be able to help you with completing the questionnaire. It should take about 10 minutes to complete the questionnaire.

Length of Study:

After you have completed the breathing tests and the questionnaires, your participation on this study will be over.

This is an investigational study. The device (called an NO breath analyzer) used in this study is FDA approved and commercially available for measuring exhaled NO levels in patients with asthma. Its use in patients with esophageal cancer is investigational. The optional SPECT scans using 99m Tc-HMPAO are an FDA approved standard imaging method for infection and/or inflammation.

Up to 150 patients (up to 93 with esophageal cancer) will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologic diagnosis of esophagus cancer.
2. For the cohort 2, patients with the pathological diagnosis of lung cancer.
3. For the cohort 3, patients with any pathological diagnosis of a thoracic malignancy.
4. Patients must sign informed consent.
5. Patients who will receive concurrent chemotherapy and radiation therapy will be undergoing PET-scan for restaging between 25 and 75 days after radio therapy.
6. For Lung Cohort, patients who will receive concurrent chemotherapy and radiation therapy or greater or equal to 3 weeks of radiation therapy alone.
7. For the Lung Cohort, participation in a PET-scan for restaging between 40-50 days after radiotherapy is required. 10 patients will receive a second PET-scan within 2-7 days as a test for reproducibility.

Exclusion Criteria:

1. Significant pleural effusion as evaluated by the attending Radiation Oncologist is excluded.
2. Patients who received thoracic radiotherapy prior to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2009-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Comparison Patient's PMRR + Mean Exhaled NO Measurement | Before starting radiation therapy (RT), after completing RT, and approximately 5 weeks later at completion of RT, and same day of restaging PET scan.
  Association between exhaled nitric oxide (NO) and PMRR (pulmonary metabolic radiation response). FDG-PET imaging (to determine PMRR) and exhaled NO assessed three times on same day of PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guerrero, MD, PhD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org